CLINICAL TRIAL: NCT01516983
Title: A Single Center, Open Label, Dose-Finding Study to Determine the Safety of Icotinib in Combination With Whole Brain Radiation Therapy For NSCLC Patients With Brain Metastases and EGFR Mutation.
Brief Title: Icotinib Combined With WBRT For NSCLC Patients With Brain Metastases and EGFR Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV04
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer; Brain Metastases
Keywords: Safety; EGFR-TKI; NSCLC; Icotinib; WBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — icotinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib+WBRT (Experimental): Standard whole brain radiotherapy plus icotinib, which is designed to administered at 5 dose according to "3+3" until disease progression or intolerable toxicity.
  Interventions: Drug: icotinib; Radiation: Whole brain radiotherapy

INTERVENTIONS:
Drug: icotinib — Level 1: Standard whole brain radiation therapy plus icotinib 125 mg Tid (375 mg per day) from day1 until disease progression or intolerable toxicity.
  Level 2: Standard whole brain radiation therapy plus icotinib 250 mg Tid (750 mg per day) from day1 until disease progression or intolerable toxicity.
  Level 3: Standard whole brain radiation therapy plus icotinib 375 mg Tid (1125 mg per day) from day1 until disease progression or intolerable toxicity.
  Level 4:Standard whole brain radiation therapy plus icotinib 500 mg Tid (1500 mg per day) from day1 until disease progression or intolerable toxicity.
  Other Names: BPI-2009, Conmana
Radiation: Whole brain radiotherapy — Whole Brain Radiation Therapy (WBRT) for total dose of 37.5Gy in 15 daily fractions beginning after Day 7.
  Other Names: RT; XRT; Radiotherapy; WBRT

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Icotinib at different dose levels in combination with whole brain radiotherapy for NSCLC patients with brain metastases and EGFR mutation.

DETAILED DESCRIPTION:
The long-term control of brain metastases becomes a clinical challenge. Whole brain radiotherapy, the standard treatment for patients with multiple brain metastases, can only bring a modest survival improvement around 3-6 months. EGFR-TKIs like icotinib with its proven activity in non-small cell lung cancer may provide clinical benefits in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small cell lung cancer (NSCLC).
* Diagnosis of brain metastases on a Gadolinium-enhanced MRI. More than 3 sites of intracranial metastases, or the longest diameter of the intracranial lesion is more than 3cm.
* Positive EGFR mutation.

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6-12 months
  All cause adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Neurological progression-free survival | 3-6 month
  All cause neurological progress or mortality
Progression-free survival | 3-6 months
  All cause progress or mortality
Overall survival | 6-12 months
  All cause mortality
Response rate | 3-6 month
Quality of life measured by FACT-L/LCS 4.0 | 1 year
Neurocognitive effects | 3-6 months
  Evaluated according to Mini-Mental Status Examination

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China